CLINICAL TRIAL: NCT04727944
Title: Evaluation of Motor-Related Beta-Activity in Relation to Naturalistic Movement in Healthy Adult Subjects
Acronym: MOBETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0843; 2021-A00042-39 (Other: ID-RCB)
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Motor Cortex; Primary Motor Cortex
Keywords: Beta burst activity; Naturalistic motor behavior; Neuroimaging techniques; electroencephalography (EEG); magnetoencephalography (MEG); magnetic resonance imaging (MRI); Reach and Grasp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEG and EEG recordings on Healthy volunteers (Experimental): All subjects can participate in experiment 1 and/or 2. All analyses are intra-subject (no analyses are between-subject).
  * Experiment 1 will test the functional role of beta bursts in naturalistic action preparation, using a combined anatomical MEG-MRI approach which will be conducted in 2 sessions.
  * Experiment 2 will study the relationship between beta bursts and naturalistic action preparation using EEG.
  Interventions: Other: Reach and grasp tasks in healthy participants using MEG technique (Experiment 1); Other: Reach and grasp tasks in healthy participants using EEG technique (Experiment 2)

INTERVENTIONS:
Other: Reach and grasp tasks in healthy participants using MEG technique (Experiment 1) — Human participants will perform reach and grasp movements to various objects (e.g. a cube, sphere, or rod) driven either by perceived action affordances, or instruction cues. A rotating carousel will be used to present subjects with various objects affording different types of grasps (e.g. a precision pinch, a whole hand 'power' grasp, or a tripod grasp).
  Prior to the experiment, subjects will be tested outside the scanner by asking them to grasp each object as they would naturally to ensure that each object elicits the expected grasp type. Subject-specific, 3D-printed head-casts will be created based on high resolution MRI scans from each subject, and worn by subjects during the MEG experiment (Experiment 1) to reduce within-session head movement associated with reaching and grasping.
  At the end of this session an experimental task is added: detection of tons in presence of multitonal masks, in order to verify how beta peaks might be generated by a stimulus auditory.
Other: Reach and grasp tasks in healthy participants using EEG technique (Experiment 2) — Experiment 2 consists of a task of reaching for and grasping several objects (e.g. a cube, sphere, or rod) ; the task used for experiment 2 is the same as that used for experiment 1. EEG signals will be measured.

SUMMARY:
The whole body's voluntary movements are controlled by the brain. One of the brain areas most involved in controlling these voluntary movements is the motor cortex and it is often viewed as the primary 'output' region of the neocortex. Motor cortical activity in the beta frequency range (13-30Hz) is a hallmark signature of healthy and pathological movement, but its behavioral relevance remains unclear. Such uncertainty confounds the development of treatments for diseases of movement which are associated with pathophysiological beta activity, including Parkinson's, therefore furthering understanding on the behavioral significance of activity in this range is now vital. Recently, it has become apparent that oscillatory beta activity actually occurs in discrete transient bursts, and that the summation of short-lasting, high-powered bursts of activity only appear to be sustained oscillations when averaged over multiple trials.

In this study we will use neurophysiological and neuroimaging techniques such as electroencephalography (EEG), magnetoencephalography (MEG), and magnetic resonance imaging (MRI). All of these techniques have been identified as non-invasive techniques. By applying these methods, we will be able to analyze beta burst activity in order to determine how beta bursts influence naturalistic motor behavior.

This project also encompasses the study of auditory and motor interactions doing an experimental task.

The aim of the project is to get a better understanding of the role of motor-related beta activity during the preparation and generation of reach and grasp actions. These findings may inform novel treatments for pathophysiological disorders characterized by aberrant beta signaling, utilizing causal manipulation of the neural circuits implicated in the generation of beta activity. This project also has expected methodological repercussions. It will make it possible to validate the use of individualized head-casts worn during MEG acquisition for the study of the cortical control of naturalistic actions, and to create new analysis tools that allow an increase in the spatial resolution of MEG data.

ELIGIBILITY:
Inclusion Criteria:

For all experiments :

* Healthy male or female
* Aged 18-40 years
* Registered with the French healthcare system
* Motivated to participate in the study
* Normal or corrected vision
* Right-handed
* Adequate knowledge of French to be able to follow directions
* Subjects must have the minimal motor ability necessary to participate in the experiment
* Subjects must be able to listen and understand the study instructions
* Subjects must be able to give written informed consent before participation
* Normal hearing

Exclusion Criteria:

For all experiments :

Subjects with characteristics incompatible with MEG/EEG and MRI :

* Claustrophobia
* Psychiatric pathology characterized including Alzheimer's disease, Parkinson's disease, multiple sclerosis (MS), or severe traumatic brain injury
* Neuropsychological disorders or cognitive impairment including schizophrenia, bipolar disorder, seizures, epilepsy, sleep disorders
* Regular use of neurodevelopment medicines (antidepressants, neuroleptics)
* Subject has a history of skin disease or skin allergies (multiple or severe)
* Subject working with metals in their professional lives
* The subject had an MRI 2 weeks prior to experiment 1
* Implanted material (any dental apparatus containing metal including or root canals or any metallic object, pacemaker, cochlear implanted in the body)
* Pregnant women or lactating women (based on self-report)
* subjects who are not able to tolerate sitting for 1 hour (the estimated length of the experiment)
* Alcohol dependence
* Subjects who, in the opinion of the investigator are not able or willing to comply with the protocol

For experiment 1:

- A head size incompatible with the use of a personalized 3D head-cast or a magnetoencephalography

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Timing of beta bursts in motor cortex, measured with MEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Timing (ms, relative to motion onset) of beta bursts in motor cortex with MEGthan the one planned is cued and must be performed.
Spatial location of beta bursts in motor cortex, measured with MEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Spatial location (mm, in a brain-centered reference frame) of beta bursts in motor cortex, measured with MEG
Timing of beta bursts in motor cortex, measured with EEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Timing (ms, relative to motion onset) of beta bursts in motor cortex with EEG
Spatial location of beta bursts in motor cortex, measured with EEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Spatial location (mm, in a brain-centered reference frame) of beta bursts in motor cortex, measured with EEG

SECONDARY OUTCOMES:
Timing of beta bursts in motor cortex, measured with MEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Timing (ms, relative to motion onset) of beta bursts in motor cortex with MEG
Spatial location of beta bursts in motor cortex, measured with MEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Spatial location (mm, in a brain-centered reference frame) of beta bursts in motor cortex, measured with MEG
Timing of beta bursts in motor cortex, measured with EEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Timing (ms, relative to motion onset) of beta bursts in motor cortex with EEG
Spatial location of beta bursts in motor cortex, measured with EEG before initiation of a movement | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Spatial location (mm, in a brain-centered reference frame) of beta bursts in motor cortex, measured with EEG
Beta amplitude, measured with MEG | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Beta amplitude (fT) in motor cortex, measured with MEG
Beta amplitude, measured with EEG | The data of subjects will be collected and analyzed through study completion an average of 2 years
  Beta amplitude (μV) in motor cortex, measured with EEG
Determine what aspects of grasp kinematics can be decoded from beta burst activity in motor cortex and related regions. | The data of subjects will be collected and analyzed through study completion an average of 2 years.
  Multivariate machine learning models which are able to predict the trajectory of arm and hand kinematics from the spatiotemporal pattern of beta bursts in motor cortex.
Within-session movement | The data of subjects will be collected and analyzed through study completion an average of 2 years.
  Movement (mm) of fiducial locations of the head-cast relative to the MEG sensors
Visual stimuli | The data of subjects will be collected and analyzed through study completion an average of 2 years.
  Comparison of synchronization, localization and waveform of beta peaks in the motor cortex in response ovisual stimuli.
Auditory stimuli | The data of subjects will be collected and analyzed through study completion an average of 2 years.
  Comparison of synchronization, localization and waveform of beta peaks in the motor cortex in response to auditory stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: James BONAIUTO, Principal Investigator — Institut des Sciences Cognitives, Marc Jeannerod, UMR 5229 CNRS
Locations (1):
- Institut des Sciences Cognitives, Marc Jeannerod, UMR 5229 CNRS, Bron, France